CLINICAL TRIAL: NCT06801184
Title: Single-center Exploratory Study of the Intestinal Microbiota in Patients Suffering of Irritable Bowel Syndrome With Predominant Constipation and Methane Production: METHANOBIOTE
Brief Title: Single-center Exploratory Study of the Intestinal Microbiota in Patients Treated for Irritable Bowel Syndrome With Predominant Constipation and Methane Production
Acronym: METHANOBIOTE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0267
Record Dates: First submitted 2025-01-13; First posted 2025-01-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: gastroenterology; microbiota; Irritable Bowel Syndrome; constipation; methano-production
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Sample:
  A peripheral venous blood sample will be collected on the day of the inclusion consultation and during the follow-up consultation at V2. These samples will be collected in 2 tubes (4 mL and 5 mL) and will be collected at the same time as the routine blood samples, which require 2 tubes (3 mL and 4 mL).
  Stool Sample:
  Approximately 1 gram of stool will be collected by the patient at home within 72 hours following the inclusion consultation and the follow-up consultation at V2, using the kits provided along with the instructions. The stools will be immediately collected into two tubes: one tube with nucleic acid preservative and one tube conservative to ensure for future metabolomic analyses. The patient will then send the sample using the pre-paid envelope included in the kit to the HCL microbiota biobank (CRB GHN) for aliquoting and storage at -80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBS patients with constipation and methane production: IBS patients with constipation and methane production
  Interventions: Biological: Plasma Sample; Biological: Stool Sample

INTERVENTIONS:
Biological: Plasma Sample — A peripheral venous blood sample will be collected on the day of the inclusion consultation and during the follow-up consultation at V2. These samples will be collected in a single2 tubes (4 mL and 5 mL)l tube and will be taken simultaneously with routine blood samples, which require 2 tubes (10 3 mL and 4 mLl).
Biological: Stool Sample — Approximately 1 gram of stool will be collected by the patient at home within 72 hours following the inclusion consultation and the follow-up consultation at V2, using the kits provided along with the instructions. The stools will be immediately collected into two tubes: one tube with nucleic acid preservative and one tube conservative to ensure for future metabolomic analyses. The patient will then send the sample using the pre-paid envelope included in the kit to the HCL microbiota biobank (CRB GHN) for aliquoting and storage at -80°C.

SUMMARY:
Irritable Bowel Syndrome (IBS), characterized by the Rome IV criteria, is a functional bowel disorder combining abdominal pain with changes in bowel habits and/or stool consistency. This condition is common, affecting 5% to 10% of the population in developed countries.

The etiology of IBS is multifactorial, involving intestinal motility disorders, visceral hypersensitivity, micro-inflammation of the intestinal mucosa, and dysbiosis. It has been demonstrated that the sub-category of IBS patients with constipation predominantly have increased amounts of Methanobrevibacter smithii, the most common methanogenic archaea found in the intestinal lumen, compared to other IBS patients.

Breath tests can evaluate methane production by the intestinal microbiota, indirectly assessing the presence and quantity of methanogenic archaea. The acronym IMO (intestinal methanogen overgrowth) defines the association of digestive symptoms (notably bloating and constipation) with a high concentration of methane in exhaled gases (≥ 10 ppm).

The links between constipation, methane production, and fecal microbiota are uncertain, necessitating further studies that could lead to precise diagnostic and treatment recommendations.

Main objective: Describe the initial composition of the fecal microbiota of constipated methano-producing IBS patients.

Secondary objectives:

2. Describe the initial composition of blood metabolites linked to the microbiota of constipated methano-producing IBS patients 3. Describe the evolution of the fecal microbiota and blood metabolites linked to the fecal microbiota during conventional therapeutic management (before and after) of constipated methano-producing IBS patients.

4. Compare the composition of the fecal microbiota before and after conventional therapeutic management of responding IBS-C patients (-30% on the IBS-SSS symptom severity score) compared to non-responding patients.

5. Evaluate the impact of Methanobrevicter smithii in the response to symptomatic treatment.

Exploratory observational single-center study (cohort follow-up) descriptive in patients with irritable bowel syndrome with constipation (IBS-C, IBS-m or IBS-U) with excessive methane production detected on a glucose breath test.

Patients will be invited to participate once the results of the breath test are known.

Please note:

In the context of this study, only two microbiota samples and 4 additional tubes and one tube of blood will be added to the usual practice. All treatments will be prescribed as part of the care and are not conditioned by the research protocol.

The primary endpoint is the analysis of the initial composition (16S rRNA gene sequencing) of the fecal microbiota of constipated methano-producing IBS patients.

The study population consists of constipated IBS patients with excessive methane production seen in the digestive functional exploration department for a breath test prescribed as part of an external procedure or a day hospital session.

A total of 40 patients will be included over 18 months, with a participation duration of 2 months +/- 2months per subject.

Patients with IBS constitute a heterogeneous population for whom only symptomatic treatment is currently offered with variable and unpredictable efficacy. Through this work, we seek to find new therapeutic axes to relieve or even treat their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from Irritable Bowel Syndrome (IBS) (abdominal pain for the past 6 months occurring on average at least 1 day per week in the last 3 months, with at least 2 of the following criteria: associated with defecation, associated with a change in stool frequency, associated with a change in stool consistency):

  1. Predominant constipation type (IBS-C): Bristol Stool Scale 1-2 ≥ 25% of the time and Bristol Stool Scale 6-7 ≤ 25% of the time
  2. Alternating diarrhea-constipation type (IBS-M): Bristol Stool Scale 1-2 25% of the time and Bristol Stool Scale 6-7 25% of the time
  3. Unspecified type: absence of sufficient criteria to meet criteria for IBS-C, IBS-D, or IBS-M.
* Patient exhibiting a high methane level (≥ 10 ppm) during a glucose breath test.
* Aged ≥ 18 years at the time of study entry.
* Patient not opposing participation in the study.

Exclusion Criteria:

* Patient who has been treated with antibiotics or probiotics in the last 3 months prior to inclusion.
* Patient suffering from diarrhea-predominant IBS (Bristol Stool Scale 6-7 ≥ 25% of the time and Bristol Stool Scale 1-2 ≤ 25% of the time).
* Patient with a history of abdominal surgery other than appendectomy and cholecystectomy.
* Patient with a history of celiac disease.
* Patient with proven inflammatory bowel disease.
* Patient with a history of colorectal cancer.
* Patient with uncontrolled hypothyroidism.
* Patient with uncontrolled diabetes.
* Pregnant or breastfeeding women.
* Patient deprived of liberty by a judicial or administrative decision.
* Adult patient under legal protection (guardianship, curators).
* Patient unable to discontinue proton pump inhibitor treatment during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with constipation-predominant irritable bowel syndrome who are methane producers suffering from constipation, attending the digestive functional explorations department for a prescribed breath test as part of an outpatient procedure or gut health workshop session.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Analysis of the initial composition (sequencing of the 16S rRNA gene) of the fecal microbiota in IBS patients with constipation and methane production. | within 2 months from the first evaluation
  16S rRNA gene sequencing is a molecular technique used to analyze the composition and diversity of microbial communities, such as those found in fecal samples. The 16S rRNA gene is a highly conserved region of bacterial and archaeal genomes, but it also contains hypervariable regions that can be used to distinguish between different species or strains.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, France